CLINICAL TRIAL: NCT02356328
Title: NovaTears® Observational Study NT-003
Brief Title: NovaTears® Eye Drops Observational Study NT-003
Status: Completed | Type: Observational
Sponsor: Novaliq GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: NT-003
Record Dates: First submitted 2015-01-21; First posted 2015-02-05 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NovaTears®
  Interventions: Device: NovaTears® Eye Drops

INTERVENTIONS:
Device: NovaTears® Eye Drops — Topical eye drops for lubrication of the ocular surface

SUMMARY:
This observational study is intended to collect outcome data from a cohort of 30 patients suffering from dry eye disease due to chronic ocular Graft-versus-Host Disease (GvHD) who are treated with the medical device NovaTears® eye drops for a duration of 11 to 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

* According to NovaTears® instruction for use
* ≥ 18 years
* Patients after an allogeneic hematopoietic stem cell transplantation with dry eye disease due to chronic ocular Graft-versus-Host Disease
* Ability and willingness to provide written Informed Consent
* Ability and willingness to participate in all examinations
* Willingness and ability to return for follow up visit

Exclusion Criteria:

* Patients with known hypersensitivity to any of the components of NovaTears®
* Patients with contact lenses, pregnancies, or who are breast feeding
* Patients with dry eye disease caused by any other known underlying systemic disease
* Patients planning an ophthalmologic surgical procedure during the course of this PMCF study
* Patients using lipid-containing or tear-film stabilizing eye drops/sprays except cyclosporin formulations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with dry eye disease due to chronic ocular GvHD
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Subjective symptom severity | 11-13 weeks
  Change in subjective symptom severity score compared to Baseline

SECONDARY OUTCOMES:
Tear-Film Break-up Time | 11 to 13 weeks
  Change in Tear Film Break-up Time (measured in seconds) compared to Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Novaliq GmbH, Study Director — Novaliq GmbH
Locations (2):
- Germany (2):
  - Department of Ophthalmology, University of Cologne, Cologne
  - University Eye Hospital Freiburg, Freiburg im Breisgau